CLINICAL TRIAL: NCT06318871
Title: A Phase 0 Pilot Study of Memory-like Natural Killer (NK) Cell Immune Therapy in Patients With Renal Cell Carcinoma or Urothelial Carcinoma
Brief Title: Memory-like Natural Killer (NK) Cell Therapy in Patients With Renal Cell Carcinoma or Urothelial Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Kidney Cancer Association (Unknown)
Responsible Party: Principal Investigator, Wenxin Xu, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-688
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Renal Carcinoma; Renal Cell Carcinoma; Urothelial Carcinoma; Chromophobe Renal Cell Carcinoma; Translocation Renal Cell Carcinoma
Keywords: Renal Carcinoma; Renal Cell Carcinoma; Advanced Clear Renal Cell Carcinoma; Urothelial Carcinoma; Translocation Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell | interventions — Cell Count; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 0: CIML NK + low dose IL-2 (Experimental): Participants will be enrolled in a staggered fashion into a 3+3 dose de-escalation design per protocol to establish a maximum tolerated dose (MTD) of CIML NK Cells. Dose will start at Dose Level 0.
  * Baseline visit.
  * Day -7: Apheresis for autologous NK cell collection.
  * Days -6 through -2: Predetermined dose of standard of care lymphodepleting chemotherapy per protocol.
  * Days 0: Predetermined dose of CIML NK Cell Therapy infusion 1x daily administered in-clinic or hospital.
  * Days 1 through 8: Low dose IL-2 every other day
  * Day 28 and then ever 2-3 months: CT/MRI/PET
  * In-clinic visit every 3 months with CT, MRI, or PET scan.
  * End of Treatment: in-clinic visit
  * Follow Up: every 4 months in-clinic, by telephone, or remotely.
  * If 2 or more out of 5 participants experience dose-limiting toxicities (DLTs), subsequent dose will be de-escalated to Dose Level -1.
  Interventions: Biological: Cytokine Induced Memory-like Natural Killer (CIML NK) Cells; Drug: Interleukin-2 (IL-2)
- Dose Level -1: CIML NK + low dose IL-2 (Experimental): Participants will complete:
  * Baseline visit.
  * Day -7: Apheresis for autologous NK cell collection.
  * Days -6 through -2: Predetermined dose of standard of care lymphodepleting chemotherapy per protocol.
  * Days 0: Predetermined dose of CIML NK Cell Therapy infusion 1x daily administered in-clinic or hospital.
  * Days 1 to 8: low dose IL-2 every other day
  * Day 28 and then ever 2-3 months: CT/MRI/PET
  * In-clinic visit every 3 months with CT, MRI, or PET scan.
  * End of Treatment: in-clinic visit
  * Follow Up: every 4 months in-clinic, by phone, or remotely.
  * If 1 or less DLTs are observed, this will be the maximum tolerated dose. If 2 or more DLTs are observed, accrual will stop.
  Interventions: Biological: Cytokine Induced Memory-like Natural Killer (CIML NK) Cells; Drug: Interleukin-2 (IL-2)

INTERVENTIONS:
Biological: Cytokine Induced Memory-like Natural Killer (CIML NK) Cells — Autologous, cytokine induced memory-like natural killer cells, via intravenous (into the vein) infusion per protocol.
  Other Names: NK Cells
Drug: Interleukin-2 (IL-2) — Interleukin-2 (aldesleukin, IL-2) will be used to support natural killer cell proliferation and activity

SUMMARY:
The goal of this research study is to establish the safety and then to explore the effectiveness of infusing the combination of cytokine-induced memory-like (CIML) natural killer (NK) cells, a type of immune cell in the blood that is collected and bathed in special proteins to help identify and treat curtained advanced cancers, combined with low dose IL-2, which is a cytokine that activates immune cells, in advanced clear cell renal cell carcinoma and urothelial carcinoma.

Names of the study therapies involved in this study are/is:

* CIML NK cell therapy (a NK cell therapy)
* IL-2 (a type of cytokine)

DETAILED DESCRIPTION:
The purpose of this research study is to obtain information on the feasibility of CIML NK cell therapy with IL-2 to treat advanced clear cell renal cell carcinoma and urothelial carcinoma. This is the first time that the specific combination of CIML NK cells and IL-2 will be given to humans.

The U.S. Food and Drug Administration (FDA) has not approved CIML NK cells post Maintenance Culture as a treatment for renal cell carcinoma or urothelial carcinoma.

The FDA has approved IL-2 as a treatment for renal cell carcinoma but the dose used will be lower than the approved dose, as IL-2 is intended to support the CIML NK cells.

This research study involves screening for eligibility, collection of natural killer (NK) cells in a process called leukapheresis, treatment visits, X-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, blood tests, urine tests, echocardiograms, electrocardiograms (ECGs), and tumor biopsies.

Participants will be in this research study for up to 5 years from the CIML NK cell infusion.

It is expected that about 10 people will take part in this research study.

This research is supported by a grant from the Kidney Cancer Association.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, advanced or metastatic clear cell renal cell carcinoma, translocation renal cell carcinoma, chromophobe renal cell carcinoma, or urothelial carcinoma. The presence of rhabdoid or sarcomatoid differentiation is permitted if a clear cell or urothelial carcinoma component is also present.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 11 (Measurement of Effect) for the evaluation of measurable disease.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of CIML NK cells in participants <18 years of age, children are excluded from this study, but would be eligible for future pediatric trials.
* Participants with clear cell RCC or UC must have progression after prior treatment failure with at least one PD-1/PD-L1 immune checkpoint inhibitor that is FDA approved for treatment of UC or RCC as of the date of informed consent.
* Patients with renal cell carcinoma should also have prior treatment failure with at least one prior VEGFR TKI, or contraindication to VEGFR TKIs as determined by the treating clinician. Patients with urothelial carcinoma should have either prior treatment failure with ≥1 prior cytotoxic chemotherapy or antibody-drug conjugate. There is no limit on the number of prior lines of therapy received.
* ECOG performance status ≤1 (Karnofsky ≥80%, see Appendix A).
* Participants must meet the following organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL
  * hemoglobin ≥8g/dL (prior transfusion permitted)
  * platelets ≥75,000/mcL
  * total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) except if secondary to Gilbert's, then < 3 x ULN
  * AST(SGOT)/ALT(SGPT) ≤3.0 × institutional ULN
  * creatinine ≤ 2.0 OR
  * glomerular filtration rate (GFR) ≥40 mL/min/1.73 m2 for participants with creatinine levels above institutional ULN.
  * oxygen saturation ≥ 90% on room air
  * left ventricular ejection fraction > 40%
  * No laboratory evidence of ongoing hemolysis in opinion of investigator
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Willing to provide blood and tissue from diagnostic biopsy
* Negative serum or urine pregnancy test at screening for women of childbearing potential. Highly effective contraception for female subjects of childbearing potential throughout the study if the risk of conception exists.
* Ability to understand and the willingness to sign a written informed consent document.
* Recipients of prior allogeneic stem cell transplantation are eligible if there is no evidence of ongoing acute or chronic graft versus host disease.

Exclusion Criteria:

* Participants who have had anti-tumor chemotherapy or other investigational agents within 2 weeks prior to enrollment(4 weeks for nitrosoureas or mitomycin C), or immunotherapy within 4 weeks prior.
* Persisting toxicity related to prior therapy (NCI CTCAE Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Prior recipients of solid organ transplantation.
* Participants who are receiving any other investigational agents.
* Participants with leptomeningeal disease are excluded from this clinical trial due to their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with treated brain metastases are eligible if imaging has shown stability over at least 4 weeks.
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn disease, are excluded from this study, as are patients with a history of active autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [Wegener's granulomatosis]) and motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis). Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or unstable cardiac arrhythmia requiring medication. Patients with rate controlled atrial fibrillation / atrial flutter on stable medical therapy are eligible.
* Other uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, or uncontrolled psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior, or other psychiatric illness/social situations that would limit compliance with study requirements, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Participants with known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of enrollment, with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other non-invasive or indolent malignancy, or cancers from which the patient has been disease-free for > 1 year after treatment with curative intent.
* No systemic corticosteroid therapy (≥ 10 mg of prednisone or equivalent dose of systemic steroids for non-autoimmune indications for at least 2 weeks prior to enrollment).
* Pregnant women are excluded from this study because of the unknown teratogenic risk of CIML NK cells and N-803 and with the potential for teratogenic or abortifacient effects by fludarabine/cyclophosphamide chemotherapy regimen. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CIML NK cells and N-803, breastfeeding should be discontinued if the mother is treated on this study. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study or 12 months after last treatment, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 12 months after completion of the last CIML NK cell and/or last N-803 administration.
* Participants with history of positive HIV testing are ineligible because of the potential for pharmacokinetic interactions with anti-retroviral agents and the treatments used in this study. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Individuals with Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive) are ineligible as they are at increased risk of lethal treatment-related hepatotoxicity.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to N-803 or other agents used in study.
* Receipt of a live vaccine within 2 weeks prior to enrollment.
* Known prior severe allergic/anaphylactic reactions to murine-based antibody therapy or iron dextran, as the CIML NK cell product contains similar reagents at end of manufacturing/infusion.
* Prior history of Grade 2 or higher hemolytic anemia (>/= 2g decrease in hemoglobin plus laboratory evidence of hemolysis) from any cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2031-07-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility Failure Rate (FFR) | Observation period up to 98 days.
  Feasibility is defined as the ability to collect cells, generate product, and administer CIML NK plus 6-day maintenance culture cells to participants. FFR is defined as the proportion pf participants that do not achieve the feasibility during the maintenance phase.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxin Xu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu